CLINICAL TRIAL: NCT02359903
Title: International Multicenter Comparative Double Blind Study of Pharmacokinetics and Safety of BCD-055 and Remicade in Patients With Ankylosing Spondylitis
Brief Title: Comparative Evaluation of Pharmacokinetics and Safety of BCD-055 and Remicade in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-055-1/ASART-1
Record Dates: First submitted 2015-01-30; First posted 2015-02-10 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab; BCD-055

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-055 group (Experimental): BCD-055 (infliximab) at a dose of 5 mg/kg, administered as a slow intravenous infusion, which will be performed on week 0, 2, 6, 14 and 22
  Interventions: Drug: Infliximab (BCD-055)
- Remicade group (Active Comparator): Remicade (infliximab) at a dose of 5 mg/kg, administered as a slow intravenous infusion, which will be performed on week 0, 2, 6, 14 and 22
  Interventions: Drug: Infliximab (Remicade)

INTERVENTIONS:
Drug: Infliximab (BCD-055) — infliximab is a chimeric monoclonal antibody against tumor necrosis factor alpha
  Other Names: Remicade; BCD-055
  Arms: BCD-055 group
Drug: Infliximab (Remicade)
  Arms: Remicade group

SUMMARY:
ASART-1 clinical study is a phase 1 study which carried out to establish the pharmacokinetic equivalence and equal safety profile of BCD-055 (infliximab manufactured by JSC BIOCAD, Russia) and Remicade when used as multiple IV infusions for the treatment of ankylosing spondylitis.

DETAILED DESCRIPTION:
ASART-1 study is the first step of clinical evaluation of infliximab biosimilar manufactured by JSC BIOCAD, Russia.The aim of this study is to establish that BCD-055 is equivalent to Remicade in terms of pharmacokinetics and safety when used by the standard regimen in patients with ankylosing spondylitis (AS).

The study will enroll 90 patients with active AS, who will be randomized into 2 groups (1:1 ratio): patients from the first group will receive BCD-055 IV at a dose 5 mg/kg on week 0, 2, 6, 14 and 22; patients from the second group will receive Remicade at the same regimen.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* active ankylosing spondylitis, which exists in patient within last 3 months
* BASDAI score > or equal to 4 points, spinal pain (by VAS) > or equal to 4 points
* history of NSAID use for the treatment of AS within last 3 months
* adequate renal and liver function
* absence of severe abnormalities in complete blood count
* consent to use adequate contraception
* ability to follow Protocol procedures

Exclusion Criteria:

* previously use of any biologic for AS treatment
* total ankylosing of the spine
* known allergy to chimeric proteins or any excipients of BCD-055/Remicade
* hepatitis B, active hepatitis C, HIV, syphilis
* known tuberculosis
* latent forms of tuberculosis
* any bacterial infection diagnosed within last month which required oral antibiotics (within last 2 weeks) or parenteral antibiotics (within last 4 weeks)
* drug or alcohol abuse
* any other disease which can affect assessments or masking some symptoms of AS (severe osteoarthrosis, nervous disorders with impairment of sensory or motor functions, another inflammatory joint disease apart from AS, etc.)
* severe uncontrolled hypertension
* chronic heart failure
* decompensated renal or liver disorders
* severe uncontrolled diabetes mellitus
* chronic obstructive lung disease, atopic bronchial asthma, angioedema in anamnesis
* any mental disorder, incl. severe depression or/and suicide thoughts/actions in anamnesis
* unstable angina pectoris
* myocardial infarction within last 12 months

Other exclusion criteria could be found in the Full Study Protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivanov Roman, PhD, Study Chair — JCS BIOCAD
Locations (6):
- Vitebsk Regional Clinical Hospital, Vitebsk, Belarus
- Russia (5):
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - Research Institute of Rheumotology, Moscow
  - Nizhegorodskaya Regional Clinical Hospital named after N.A. Semashko, N.Novgorod
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg
  - Local hospital at the station Smolensk OAO RZD, Smolensk

RESULTS

PARTICIPANT FLOW:
Groups:
- Remicade Group: Remicade (infliximab) at a dose of 5 mg/kg, administered as a slow intravenous infusion, which will be performed on week 0, 2, 6, 14 and 22
  Infliximab (Remicade)
Period: Overall Study
Arm/Group | BCD-055 Group | Remicade Group
Started | 45 | 45
Completed | 45 | 43
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: All patients who received at least 1 injection of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-055 Group | Remicade Group | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [32 to 51] | 38 [35 to 55] | 38 [33 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 336 Hours After the Single Infusion of BCD-055/Remicade
Time Frame: 2 weeks
Population: Patients who received at least 1 injection. From BCD-055 group 1 patient was excluded because of violation of timing of blood collection. From Remicade group 2 patients were excluded due to AE/SAE.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Arm/Group | BCD-055 Group | Remicade Group
Number analyzed (Participants) | 44 | 43
(ng/ml)*hour | 26282582 [21094742 to 32296361] | 25914888 [20105020 to 32661812]

2. Secondary Outcome: Maximum Concentration of Infliximab After the Single Infusion of BCD-055/Remicade
Description: Patients who received at least 1 injection. From BCD-055 group 1 patient was excluded because of violation of timing of blood collection. From Remicade group 2 patients were excluded due to AE/SAE.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | BCD-055 Group | Remicade Group
Number analyzed (Participants) | 44 | 43
ng/ml | 174638 [139415 to 239141] | 195434 [134622 to 257656]

3. Secondary Outcome: Time of Maximum Concentration of Infliximab After the Single Infusion of BCD-055/Remicade
Time Frame: 2 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Maximum Concentration of Infliximab After the 1st, 2nd, 3rd, 4th and 5th Infusion of BCD-055/Remicade
Time Frame: 28 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Minimum Concentration of Infliximab After the 1st, 2nd, 3rd, 4th and 5th Infusion of BCD-055/Remicade
Time Frame: 28 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Time of Maximum Concentration of Infliximab After the1st, 2nd, 3rd, 4th and 5th Infusion of BCD-055/Remicade
Time Frame: 28 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Half Life of Infliximab After the 1st and 5th Infusion of BCD-055/Remicade
Time Frame: 2 weeks / 28 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Average Concentration of Infliximab at Steady State Phase
Time Frame: 28 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Patients in Each Group Achieving ASAS20
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Percentage of Patients in Each Group Achieving ASAS40
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Mean Change of BASDAI Score Compared With Baseline
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Mean Change of BASMI Score Compared With Baseline
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Mean Change of BASFI Score Compared With Baseline
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Mean Change of MASES Score Compared With Baseline
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Mean Change of SF36 Score Compared With Baseline
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Mean Change of Chest Expansion Compared With Baseline
Time Frame: 14 weeks / 30 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Frequency of AE/SAE After the Single Infusion of BCD-055/Remicade
Time Frame: 2 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Total Frequency of AE/SAE Within the Whole Time of the Study
Time Frame: 30 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Total Frequency of Grade 3-4 Laboratory Abnormalities Within the Whole Time of the Study
Time Frame: 30 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Percentage of Patients in Whom Bind or Neutralizing Antibodies to Infliximab Were Detected
Time Frame: screening / 14 weeks / 30 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Frequency of Early Withdrawal Due to AE/SAE
Time Frame: 30 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Maximum Concentration at Steady State
Time Frame: 28 weeks
Reporting Status: Not Posted, anticipated posting 2016-12

23. Other Pre Specified Outcome: Area Under the Plasma Concentration-time Curve at Steady State Phase
Time Frame: 28 weeks
Reporting Status: Not Posted, anticipated posting 2016-12

ADVERSE EVENTS:
Arm/Group | BCD-055 Group | Remicade Group
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/45
Other Adverse Events (participants affected / at risk) | 4/45 | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-055 Group (N=45) | Remicade Group (N=45)
Collapse (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-055 Group (N=45) | Remicade Group (N=45)
Arterial hypertension (Blood and lymphatic system disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No